CLINICAL TRIAL: NCT06014840
Title: Early Diagnosis and Treatment of Undiagnosed COPD or Asthma: The UCAP 2 Trial - Pilot Study
Brief Title: The UCAP 2 Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started, no participants were enrolled. The protocol was significantly changed and current described study was abandoned.
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023
Record Dates: First submitted 2023-07-31; First posted 2023-08-28 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: COPD; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — Restraint, Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early diagnosis and treatment of COPD or Asthma (Active Comparator): Treatment strategy using evidence-based guidelines for asthma or COPD provided to participant on the day of randomization
  Interventions: Other: Assessment and Treatment provided to participant by a respirologist using evidence-based guidelines for asthma or COPD
- Delayed diagnosis and treatment of COPD or Asthma (Other): Treatment strategy using evidence-based guidelines for asthma or COPD provided to participant at 12 weeks.
  Interventions: Other: Assessment and Treatment provided to participant by a respirologist using evidence-based guidelines for asthma or COPD

INTERVENTIONS:
Other: Assessment and Treatment provided to participant by a respirologist using evidence-based guidelines for asthma or COPD — Assessment and Treatment provided to participant by a respirologist using evidence-based guidelines for asthma or COPD

SUMMARY:
Our research group has found that Canadians with undiagnosed asthma or chronic obstructive pulmonary disease (COPD) have increased respiratory symptoms and worse health-related quality of life.

The investigators recently developed and validated an on-line questionnaire to accurately identify these symptomatic, undiagnosed individuals.

The investigators will advertise in the community asking individuals to complete the on-line questionnaire at home, at their leisure, to determine if they are at risk of asthma or COPD. Those at risk will be invited to participate in our randomized, controlled clinical trial to determine if guidelines-based treatment of newly discovered undiagnosed asthma or COPD will improve their quality of life and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals at least 18 years old
* Individuals must be symptomatic with respiratory symptoms
* Individuals must complete the UCAP-Q questionnaire and score a ≥ 6% probability of having either asthma or COPD.
* Individuals who have given written informed consent to participate in this trial in accordance with local regulations;
* Individual must be able to perform pre and post bronchodilator spirometry to measure lung function

Additional Inclusion Criteria for the Randomized Controlled Trial (RCT):

* Individuals who have undiagnosed airflow obstruction (i.e. Asthma will be diagnosed in subjects with airflow obstruction whose forced expiratory volume in 1 second (FEV1) improves by > 12% and 200 ml after bronchodilator and COPD will be diagnosed in subjects who do not have a significant bronchodilator response and who exhibit persistent airflow obstruction post bronchodilator) will be asked to participate in the RCT.

Exclusion Criteria:

* Individuals who report a previous diagnosis of asthma, COPD, history of lung cancer, bronchiectasis, interstitial lung disease, cystic fibrosis or other significant diagnosed lung disease.
* Individuals currently under the care of a respirologist
* Individuals currently using inhaled corticosteroids or long-acting bronchodilators.
* Individuals with history of myocardial infarction, stroke, aortic or cerebral aneurysm, or detached retina or eye surgery within the past 3 months (spirometry is contraindicated)
* Individuals who are in the third trimester of pregnancy
* Individuals involved in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in disease-specific quality of life quantified using the St. George's Respiratory Questionnaire (SGRQ). | 12 weeks
  The change in disease-specific quality of life will be expressed as the total St. George's Respiratory Questionnaire score at 12 weeks minus the score on the day of randomization. This questionnaire includes 3 domains: symptoms (distress caused by specific respiratory symptoms); activity (physical activities that cause or are limited by breathlessness); and impact (social and psychological effects of the respiratory disease). A total change of - 4 points in the SGRQ total score has been established as the minimal clinically important difference (MCID) for this questionnaire. Higher scores indicate poor health status.

SECONDARY OUTCOMES:
Change in dyspnea as assessed by The Baseline and Transitional Dyspnea Indexes | 12 weeks
  The baseline dyspnea index (BDI) is used to rate the severity of dyspnea at a single point in time and the transition dyspnea index (TDI) is used to assess changes from that baseline. The change in dyspnea will be expressed as the total score at 12 weeks minus the score on the day of randomization. A total change of more than 1 point in the score has been established as the minimal clinically important difference (MCID) for this questionnaire.
Changes in overall respiratory symptoms (including cough, sputum and dyspnea) will be assessed using the COPD Assessment Test (CAT) | 12 weeks
  The change in overall respiratory symptom burden will be expressed as the total score of the COPD Assessment Test at 12 weeks minus the score on the day of randomization. A total change of 2 points in the CAT total score has been established as the minimal clinically important difference (MCID) for this questionnaire. Higher scores indicate higher burden.
Changes in absenteeism and presenteeism as assessed by the Work Productivity and Activity Impairment Questionnaire (WPAI) | 12 weeks
  The change in absenteeism and presenteeism will be assessed over the 12 week study period. Higher scores indicate greater impairment in work productivity and daily activities.
Quality of life changes as assessed by the 36-Item Short Form Health Survey (SF-36) Health Survey Questionnaire | 12 weeks
  The change in general health status will be expressed as the total score of the SF-36 Health Survey Questionnaire at 12 weeks minus the score on the day of randomization. A total change of 8-10 points in the SF-36 has been established as the minimal clinically important difference (MCID) for this questionnaire. Higher scores indicate better health status.
Changes in forced expiratory volume in one second (FEV1) measured in litres (L) using pre bronchodilator spirometry testing and post bronchodilator spirometry testing. | 12 weeks
  The change will be expressed as the mean change in the FEV1 measurements at 12 weeks in comparison to the lung function measurements on the day of randomization.
Differences between groups in patient-initiated healthcare utilization events for respiratory illness over the 12-week trial period. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Vandemheen, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital General Campus, Ottawa, Ontario, Canada